CLINICAL TRIAL: NCT00050570
Title: Interventions to Reduce Eating Disorder Risk Factors
Brief Title: Reducing Eating Disorder Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Craig Barr Taylor, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH060453 (NIH); R01MH060453 (NIH); DSIR CT-P
Record Dates: First submitted 2002-12-16; First posted 2002-12-17 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

ARMS (2):
- Intervention (Experimental): An 8-week, Internet- based, structured cognitive- behavioral program combined with an online, asynchronous, moderated discussion group.
  Interventions: Behavioral: Web-based intervention to reduce eating disorder risk factors
- Control (No Intervention): The waitlist control group was only contacted at the time of assessments and was offered the intervention at the end of the study, after the 2-year follow-up assessment was completed.

INTERVENTIONS:
Behavioral: Web-based intervention to reduce eating disorder risk factors
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether a web-based program is effective in reducing the incidence of eating disorders in college women who are at high risk for developing an eating disorder.

DETAILED DESCRIPTION:
Female college students who use unhealthy weight control methods and have body image concerns may be at risk for developing an eating disorder. Developing and evaluating interventions to reduce eating disorders in high-risk populations is of great public health importance.

Participants are randomly assigned to either join a web-based risk-reduction program or receive no intervention. The 9-week risk-reduction program focuses on reducing body image and weight/shape concerns, identifying the risks of eating disorders, and increasing healthy weight regulation practices. The program includes weekly readings, writing assignments, and participation in a moderated electronic discussion group. Changes in body mass index (BMI) and the occurrence of major stressors and psychiatric events are assessed to determine their impact on the incidence of eating disorders. One-year incidence of eating disorders is determined by a diagnostic interview, and follow up may continue for up to 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* College students at risk for developing an eating disorder

Exclusion Criteria:

* Suicidal or other severe psychopathology
* Alcohol or drug abuse
* Body mass index (BMI) < 18 or > 32
* Current diagnosis of anorexia nervosa, binge eating disorder, or bulimia nervosa and have been in treatment within the past 6 months

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2001-02; Primary Completion 2012-04-30 (Actual); Study Completion 2012-04-30 (Actual)

PRIMARY OUTCOMES:
Onset of an eating disorder | 2 years
  The main outcome is the onset of an eating disorder, as defined by DSM-IV

SECONDARY OUTCOMES:
Change in eating disorder behaviors | 2 years
  Eating disorder behaviors as measured by the Eating Disorder Examination. We will also measure attitudes related to eating disorder onset risk

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Dept. of Psychiatry and Behavioral Sciences, Stanford, California, United States